CLINICAL TRIAL: NCT01093833
Title: A Comparison Study of Prototype Continuous Glucose Sensors in the Intradermal and Subcutaneous Spaces
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BDT-08-CGM-02
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
Keywords: Diabetes; Type 1 diabetes; Type 2 diabetes; Diabetes mellitus; Blood glucose; Continuous blood glucose monitoring; CGM
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous Glucose Monitoring (Experimental): Each subject will participate in one experimental intervention. Blood glucose will be measured with the BD continuous glucose monitor (BD CGM), with the Medtronic Guardian CGM and the YSI Glucose Analyzer as controls for 12-14 hours.
  Interventions: Device: BD Continuous glucose monitor (BD CGM); Device: YSI Glucose Analyzer; Device: Medtronic Guardian CGM

INTERVENTIONS:
Device: BD Continuous glucose monitor (BD CGM) — Continuous glucose monitoring for 12-14 hours
  Other Names: MiniMed Guardian CGM
Device: YSI Glucose Analyzer — Continuous glucose monitoring for 12-14 hours
Device: Medtronic Guardian CGM — Continuous glucose monitoring for 12-14 hours

SUMMARY:
The purpose of this study is to compare two continuous glucose sensors, one placed subcutaneous (under the skin) and one placed intradermal (in the skin) over 12-14 hours.

DETAILED DESCRIPTION:
This was a single site, non-randomized study. The study consisted of a screening visit (Visit 1), during which the subject was consented and the inclusion and exclusion criteria confirmed, an experimental intervention (Visit 2) and a follow-up visit (Visit 3). The experimental intervention was based on an initial glucose clamp involving a basal intravenous (IV) insulin infusion and IV insulin boluses plus IV glucose infusion / IV glucose boluses as required to maintain euglycemic, hypoglycemic and hyperglycemic plateaus respectively in 41 subjects with Type 1 or Type 2 Diabetes. At the end of hour five of the study the glucose clamp was discontinued and subjects given a standardized meal to stimulate a hyperglycemic excursion

Each subject participated in one experimental intervention. During the glucose clamp intervention, the subject's blood glucose was continuously monitored either by means of the Biostator or by frequent venous blood glucose measurements based on a standard lab method (YSI STAT2300 analyzer), and measured by means of the BD Technologies test devices, and the Medtronic Guardian CGM. Once the clamp was discontinued the Biostator was discontinued as well. During the unclamped period and meal the subjects BG was monitored via the YSI Glucose Analyzer, the BD CGM sensor and the Medtronic Guardian CGM.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male and female subjects with Type 1 or Type 2 diabetes mellitus
* Signed informed consent
* Age between 18 and 65 years, inclusive
* Body mass index between 19 and 30 kg/m², inclusive
* HbA1c < 11 %

Exclusion Criteria:

* Uncontrolled arterial hypertension (diastolic blood pressure >90 mm Hg and/or systolic blood pressure >160 mm Hg)
* Impaired hepatic function measured as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ three times the upper reference limit
* Impaired renal function measured as creatinine > 1.2 times above the upper limit of normal.
* Severe acute diseases, i.e. cardiac, pulmonary, gastrointestinal, hepatic, neurologic, or infectious that might interfere with the performance of this study, as judged by the Investigator.
* Severe chronic diseases, as judged by the investigator other than Type 1 Diabetes
* Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device.
* Known microvascular (diabetic) complications (other than diabetic non-proliferative retinopathy), such as e.g. history of laser coagulation, proliferative diabetic retinopathy, known diabetic nephropathy or neuropathy requiring treatment
* Positive serology for Hepatitis B, Hepatitis C or HIV
* Pregnancy, breast-feeding or intention of becoming pregnant or not using adequate contraceptive measures.
* Known current or recent alcohol or drug abuse
* Blood donation of more than 500 ml within the last three months
* Anticoagulant therapy
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
* Previous participation in a study involving the GBP-based sensor
* Has taken more than 4000 mg or more of acetaminophen within the past 24 hours (i.e. 13 or more regular strength or 8 or more extra strength Tylenol in the past 24 hours)
* Any skin condition that may be judged to have affect on study ( e.g., bad sunburn, pre-existing dermatitis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 12-14 hours

CONTACTS AND LOCATIONS:
Overall Officials: Morrow Linda, MD, Principal Investigator — Profil Insitute for Clinical Research
Locations (1):
- Profil Institute for Clinical Research Inc, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Judge K, Morrow L, Lastovich AG, Kurisko D, Keith SC, Hartsell J, Roberts B, McVey E, Weidemaier K, Win K, Hompesch M. Continuous glucose monitoring using a novel glucose/galactose binding protein: results of a 12-hour feasibility study with the becton dickinson glucose/galactose binding protein sensor. Diabetes Technol Ther. 2011 Mar;13(3):309-17. doi: 10.1089/dia.2010.0130. Epub 2011 Feb 7. PMID 21299393